CLINICAL TRIAL: NCT01813071
Title: A Randomized, Double-Blinded, Placebo-controlled, Dose-Escalation, Age-Descending Study to Assess the Safety and Tolerability of Live Attenuated, Oral Shigella WRSS1 (Walter Reed S. Sonnei) Vaccine in Bangladeshi Adults and Children
Brief Title: Safety Study of Live Attenuated Oral Shigella (WRSS1) Vaccine in Bangladeshi Adults and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC 008; PR-12054 (Other: International Centre for Diarrhoeal Disease Research)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Diarrhea
Keywords: Enterobacteriaceae Infections; Gram-Negative Bacterial Infections; Bacterial Infections; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Shigellosis
MeSH Terms: conditions — Diarrhea; Enterobacteriaceae Infections; Gram-Negative Bacterial Infections; Bacterial Infections; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Part A (Adults): Cohort A1 (Experimental): One oral dose of ~3x10^4 cfu WRSS1(10 participants) or placebo (3 participants)
  Interventions: Biological: WRSS1
- Part A (Adults): Cohort A2 (Experimental): Three oral doses of ~3x10^5 cfu WRSS1(10 participants) or placebo (3 participants)
  Interventions: Biological: WRSS1
- Part A (Adults): Cohort A3 (Experimental): Three oral doses of ~3x10^6 cfu WRSS1(10 participants) or placebo (3 participants)
  Interventions: Biological: WRSS1
- Part B (Children): Cohort B1 (Experimental): One oral dose of ~3x10^3 cfu WRSS1(12 participants) or placebo (4 participants)
  Interventions: Biological: WRSS1
- Part B (Children): Cohort B2 (Experimental): Three oral doses of ~3x10^4 cfu WRSS1(12 participants) or placebo (4 participants)
  Interventions: Biological: WRSS1
- Part B (Children): Cohort B3 (Experimental): Three oral doses of ~3x10^5 cfu WRSS1(12 participants) or placebo (4 participants)
  Interventions: Biological: WRSS1
- Part B (Children): Cohort B4 (Experimental): Three oral doses of ~3x10^6 cfu WRSS1(12 participants) or placebo (4 participants)
  Interventions: Biological: WRSS1

INTERVENTIONS:
Biological: WRSS1

SUMMARY:
This is a research study about an experimental (investigational) oral Shigella sonnei - Walter Reed S. sonnei (WRSS1). WRSS1 is a live vaccine that is being made to prevent disease from Shigella, which causes bloody, watery diarrhea. Infants and children living in developing countries experience the greatest consequences of this disease. The purpose of this study is to find a dose of the vaccine that is safe, tolerable, and develops an immune response. About 39 healthy adults, ages 18-39, and 48 healthy children, ages 5-9, will participate in this study. Once the vaccine is proven safe and tolerable in adults, then it will be tested in the children. This study will require volunteers to stay in the research facility for several nights for the first dose; they will not be required to stay overnight for the second and third doses. Participants will be assigned to receive 1 of 3 vaccine dose levels by mouth. Study procedures include: stool samples, blood samples and documenting side effects. Participants will be involved in study related procedures for about 8 months.

DETAILED DESCRIPTION:
This is a single site, double-blind, randomized, placebo-controlled, dose-escalation, age-descending study that will start testing the vaccine in healthy adults and move subsequently into school-age children. The study is designed as 2 parts, each part comprising 3 cohorts. The cohort receiving the lowest dose in Parts A and B will receive only one administration of vaccine or placebo; the subsequent two higher dose cohorts in Parts A and B will receive three administrations of vaccine or placebo. In each cohort, the first dose and immediate safety evaluation will be conducted at the International Centre for Diarrhoeal Disease Research (icddr,b) Inpatient Unit, where the participants will be admitted for observation for 72 hours. Follow-up visits for participants in A1 and B1 will take place on an outpatient basis at the Mirpur, Bangladesh (Mirpur) Field Office. Second and third vaccinations within A2, A3, B2, and B3 cohorts and all follow-up visits will take place on an outpatient basis at the Mirpur Field Office. Before enrolling participants in subsequent cohorts to receive a higher vaccine dose, or to move to the lower age group, the safety data from the previous cohort(s) (through Study Day 7) will be evaluated and reviewed by the Internal Protocol Safety Team (IPST) comprised of the study physician, the Medical Monitor from GVK Biosciences (GVK), the principal investigator, and the Medical Monitor from PATH Vaccine Solutions (PVS). Upon completion of the last adult cohort, the Data Safety Monitoring Board (DSMB -an advisory body to the Ethical Review Committee) will convene to review the cumulative safety data and IPST recommendation, and determine whether to proceed to Part B (children). Adverse events (AE)s will be graded according to standardized criteria. The immunogenicity outcome measures of interest include serum immunoglobulin G (IgG) and immunoglobulin A (IgA) antibodies by Antibodies in Lymphocyte Supernatant (ALS) assay against S. sonnei2a lipopolysaccharide (LPS), shedding profile of WRSS1, and vaccine-specific mucosal IgA responses.

The proposed study builds upon successful preliminary observations with this vaccine in the US, Israel and Thailand. While secondary objectives include studying the immunogenicity of the WRSS1 vaccine, the primary goal of the current trial is to establish a clear safety profile for the WRSS1 vaccine in adults and children 5-9 years old.The primary objective of the study is to evaluate the safety and tolerability of the vaccine; the secondary objective is to evaluate vaccine immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults from 18-39 years old, inclusive
* General good health as determined by the screening evaluation no greater than 30 days before admission
* Properly informed about the study, able to understand it and sign the informed consent form
* Normal bowel habits (< 3 grade 1 or 2 stools each day; ≥ 1 grade 1 or 2 stools every 2 days)
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Available for the entire period of the study and reachable by study staff throughout the entire follow-up period
* Females of childbearing potential who are willing to take a serum pregnancy test at screening and urine pregnancy tests before each vaccination. Pregnancy tests must be negative before each vaccination. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is also acceptable.
* Signed Informed Consent

Exclusion Criteria:

* Presence of a significant medical or psychiatric condition that in the opinion of the Investigator precludes participation in the study
* Known infection with Hepatitis C or Human Immunodeficiency Virus (HIV)
* History of congenital abdominal disorders, intussusception, abdominal surgery or any other congenital disorder.
* Participation in research involving another investigational product (defined as receipt of investigational product) 30 days before planned date of first vaccination or concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational product
* Clinically significant abnormalities on physical examination
* Clinically significant abnormalities in screening hematology, serum chemistry, or urinalysis as determined by the PI or the PI in consultation with the Study Physician
* History of febrile illness within 48 hours prior to vaccination
* Known or suspected impairment of immunological function based on medical history and physical examination
* Prior receipt of any Shigella vaccine
* Fever at the time of immunization. Fever is defined as a temperature ≥ 37.5 degrees Celsius (99.5 degrees Fahrenheit) on axillary, oral, or tympanic measurement
* Clinical evidence of active gastrointestinal illness
* Prior receipt of a blood transfusion or blood products, including immunoglobulins
* Presence of any significant systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would endanger the participant's health or is likely to result in non-conformance to the protocol.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment
* Evidence of current excessive alcohol consumption
* Evidence of current illicit drug use or drug dependence
* Current use of iron or zinc supplements within the past 7 days; current use of antacids (Histamine H2-receptor antagonists (H2 blockers), Omeprazole, over the counter (OTC) agents) or immunosuppressive drug
* Allergy to quinolone, sulfa, and penicillin classes of antibiotics
* History of any of the following conditions within the past 10 years:

  1. Arthritis (two or more episodes of joint pain and swelling)
  2. Gastrointestinal disease (diagnosed by a doctor as having irritable bowel disease, Crohn's disease, ulcerative colitis (biopsy confirmed), celiac disease, stomach or intestinal ulcers
  3. Dyspepsia (indigestion or heartburn requiring medication more than once per week)
  4. History of gallbladder disease
  5. History of chronic heart disease
* Any conditions which, in the opinion of the investigator, might jeopardize the safety of study participants or interfere with the evaluation of the study objectives
* Receipt of antimicrobial drugs for any reason or a fever ≥ 38 degrees Celsius within 7 days before vaccination
* History of diarrhea during the 7 days before vaccination.
* Has any household member(s) who is immunocompromised or under the age of 2 years old.

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubhana Raqib, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sarker P, Mily A, Ara A, Haque F, Maier N, Wierzba TF, Walker RI, Venkatesan MM, Raqib R. Functional Antibodies and Innate Immune Responses to WRSS1, a Live Oral Shigella sonnei Vaccine Candidate, in Bangladeshi Adults and Children. J Infect Dis. 2021 Dec 20;224(12 Suppl 2):S829-S839. doi: 10.1093/infdis/jiab395. PMID 34374425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in general good health were recruited, screened and consented at the icddr,b Dhaka in Bangladesh. Final eligibility was determined by fulfillment of all the inclusion and absence of any of the exclusion criteria. Adults were enrolled August 23, 2013 to November 10, 2013 and children were enrolled April 27, 2014 to August 9, 2015.
Groups:
- Part A (Adults): Cohort A1: One oral dose of ~3x10^4 cfu WRSS1
- Part A (Adults): Cohort A2; Part B (Children): Cohort B3: Three oral doses of ~3x10^5 cfu WRSS1
- Part A (Adults): Cohort A3; Part B (Children): Cohort B4: Three oral doses of ~3x10^6 cfu WRSS1
- Part A (Adults): Placebo; Part B (Children): Placebo: One or Three oral doses of Placebo
- Part B (Children): Cohort B1: One oral dose of ~3x10^3 cfu WRSS1
- Part B (Children): Cohort B2: Three oral doses of ~3x10^4 cfu WRSS1
Period: Overall Study
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
Started | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16
Completed | 10 | 10 | 10 | 9 | 11 | 5 | 9 | 7 | 13
Not Completed | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 5 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Met inc/exc criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Additional row added to stratify participants by 'adults' and 'children' and give totals for each.
  years
    Part A Adults: number analyzed (Participants) | 10 | 10 | 10 | 9 | 0 | 0 | 0 | 0 | 0 | 39
    Part A Adults | 25.7 (5.23) | 28.1 (5.51) | 27.0 (2.67) | 27.4 (5.34) |  |  |  |  |  | 27.1 (4.71)
    Part B Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 16 | 64
    Part B Children |  |  |  |  | 6.3 (0.98) | 6.6 (1.16) | 6.0 (0.85) | 6.3 (0.97) | 6.6 (1.02) | 6.4 (1.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 4 | 8 | 8 | 9 | 5 | 12 | 63
  Male | 5 | 5 | 3 | 5 | 4 | 4 | 3 | 7 | 4 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bangladesh | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16 | 103
Height (cm) [Mean (Standard Deviation); unit: centimeters] — Population: Additional row added to stratify participants by 'adults' and 'children' and give totals for each.
  centimeters
    Part A Adults: number analyzed (Participants) | 10 | 10 | 10 | 9 | 0 | 0 | 0 | 0 | 0 | 39
    Part A Adults | 160.7 (10.75) | 160.1 (9.47) | 157.0 (6.36) | 159.2 (10.07) |  |  |  |  |  | 159.3 (9.03)
    Part B Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 16 | 64
    Part B Children |  |  |  |  | 116.4 (4.66) | 116.4 (8.32) | 115.0 (4.86) | 121.0 (6.74) | 119.4 (7.91) | 117.8 (6.90)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] — Population: Additional row added to stratify participants by 'adults' and 'children' and give totals for each
  kilograms
    Part A (Adults): number analyzed (Participants) | 10 | 10 | 10 | 9 | 0 | 0 | 0 | 0 | 0 | 39
    Part A (Adults) | 67.3 (13.98) | 58.1 (11.52) | 54.5 (8.43) | 56.4 (11.52) |  |  |  |  |  | 59.2 (12.16)
    Part B (Children): number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 16 | 64
    Part B (Children) |  |  |  |  | 19.7 (1.64) | 20.5 (4.09) | 21.3 (4.26) | 22.9 (4.62) | 21.0 (3.81) | 21.1 (3.85)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events (SAEs)
Description: Based on maximum severity per participant over all serious adverse events (SAEs) within 6 months of any vaccination. A Serious Adverse Event, including serious suspected adverse reaction or serious adverse reaction as determined by the Investigator or the sponsor, was any event that results in any of the following outcomes: Inpatient hospitalization or prolongation of existing hospitalization , life-threatening AE that in the opinion of the investigator or sponsor put the participant at immediate risk of death, persistent or significant incapacity or substantial disruption, congenital abnormality or birth defect, a medically important event that may have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed or death.
Time Frame: Day -1(admission day) through 6 months (Day 224 +/- 14 days) after the third vaccination for Cohorts A2,A3, B2, B3, B4, and after the first vaccination (Day 168 +/- 14 days) for Cohorts A1 and B1.
Population: All participants who had been exposed to at least one dose of study product were included in the primary analysis for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1

2. Primary Outcome: Number and Percentage of Participants With Any Non-serious Unsolicited Adverse Events
Description: Based on subject count over all non-serious adverse events. An Adverse event was defined as any untoward medical occurrence in humans, whether or not considered drug related, that occurred during the conduct of a clinical trial. Any change in clinical status, ECGs, routine labs, x-rays, physical examinations, etc., that was considered clinically significant by the study investigator, was considered an AE. This definition also included an exacerbation or worsening of pre-existing conditions or events, inter-current illnesses, injuries, or vaccine or drug interaction, or worsening of abnormal clinical laboratory values. All AEs were assessed by the clinician using a protocol defined grading system.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16
Participants | 8 | 7 | 8 | 6 | 10 | 9 | 9 | 12 | 12

3. Primary Outcome: Number and Percentage of Participants With Solicited Systemic and Intestinal Reactions
Description: Maximum severity per participant of any systemic or any gastrointestinal reactogenicity recorded within 7 days of any vaccination is reported. Solicited Systemic reactogenicity events assessed included fever, headache, malaise, generalized myalgia, arthralgia, chills, reactive arthritis and decreased appetite. Intestinal solicited reactogenicity events assessed included abdominal cramps, abdominal pain, nausea, vomiting, loose stool, diarrhea, dysentery, bloating, excess flatulence and constipation. Diarrhea and dysentery were assessed both during inpatient (first three day period post-vaccination) and outpatient ( post-vaccination days 4-7) periods post-vaccination 1. Vaccinations 2 and 3 did not have an inpatient admission period for any participants. Diarrhea severity was determined on the basis of stool number, grading and stool weight during the inpatient period and by stool number and grading only during the outpatient period.
Time Frame: Day 0 through Day 7 after any vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16
Participants
  Any Systemic Reactogenicity | 2 | 1 | 6 | 4 | 0 | 3 | 0 | 4 | 2
  Any Gastrointestinal Reactogenicity | 2 | 4 | 7 | 4 | 2 | 4 | 3 | 6 | 2

4. Primary Outcome: Number and Percentage of Participants With Any Unsolicited AEs and SAEs Judged as Having a Reasonable Possibility That the Study Product Caused the Event
Description: Adverse event (AE) was defined as any untoward medical occurrence in humans, whether or not considered drug related, that occurs during the conduct of a clinical trial. A Serious Adverse Event (SAE) , including serious suspected adverse reaction or serious adverse reaction as determined by the Investigator or the sponsor, was any event that results in any of the following outcomes: Inpatient hospitalization or prolongation of existing hospitalization , life-threatening AE that in the opinion of the investigator or sponsor put the participant at immediate risk of death, persistent or significant incapacity or substantial disruption, congenital abnormality or birth defect, a medically important event that may have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed or death. Causality of the AE/SAE to the study drug was assessed by the Investigator as reasonable possibility that the study product caused the reported event.
Time Frame: SAEs at any time and AEs after any vaccination until Day 168 (Cohort A1, B1) and Day 224 (all other Cohorts).
Population: All participants who had been exposed to at least one dose of study product were included in the primary analysis for safety. Adult Cohort A1 and Child Cohort B1 only received a single dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 12 | 12 | 12 | 12 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Immunoglobulin A (IgA) Antibodies in Antibody Titers in Lymphocyte Supernatant (ALS)
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific immunoglobulin A (IgA) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and a novel composition comprising invasin proteins and LPS from gram-negative bacteria (Invaplex) using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgA responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom research blood was collected and analyzed. Adult Cohort A1 and Child Cohort B1 received a single dose of study vaccine and had research blood collected only on Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 3 | 6 | 7 | 0 | 0 | 0 | 1 | 3
  LPS | 0 | 3 | 7 | 7 | 0 | 0 | 0 | 1 | 3

6. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in ALS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgA (immunoglobulin A) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgA responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 35
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 2 | 4 | 1 |  | 0 | 1 | 3
  LPS | 0 |  | 2 | 4 | 0 |  | 0 | 1 | 2

7. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in ALS
Description: as for outcome 6
Time Frame: Day 63
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 7 | 11 | 10
Participants
  Invaplex | 0 |  | 1 | 3 | 0 |  | 0 | 0 | 3
  LPS | 0 |  | 1 | 5 | 0 |  | 0 | 1 | 3

8. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in ALS
Description: as for outcome 6
Time Frame: At any time (Day 7 to Day 63)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 3 | 7 | 8 | 1 | 0 | 0 | 2 | 4
  LPS | 0 | 3 | 7 | 8 | 0 | 0 | 0 | 3 | 4

9. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Immunoglobulin G (IgG ) IgG Antibodies in ALS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific immunoglobulin G (IgG ) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgG responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 3 | 3 | 4 | 0 | 1 | 0 | 1 | 1
  LPS | 0 | 2 | 6 | 7 | 0 | 0 | 0 | 1 | 4

10. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in ALS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgG (immunoglobulin G) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgG responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 35
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 1 |  | 3 | 1 | 1 |  | 1 | 3 | 2
  LPS | 0 |  | 4 | 6 | 0 |  | 0 | 1 | 2

11. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in ALS: Invaplex
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgG (immunoglobulin G) antibody responses to S. sonnei 2a Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine Invaplex-specific IgG responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 63
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 7 | 10 | 10
Participants | 1 |  | 2 | 2 | 0 |  | 0 | 0 | 4

12. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in ALS: Lipopolysaccharide (LPS)
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgG (immunoglobulin G) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS-specific IgG responses from circulating lymphocytes. Proportion of participants with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 63
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 7 | 11 | 10
Participants | 0 |  | 2 | 6 | 0 |  | 0 | 0 | 3

13. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in ALS
Description: as for outcome 10
Time Frame: At any time (Day 7 to Day 63)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 3 | 5 | 5 | 1 | 1 | 1 | 3 | 5
  LPS | 0 | 2 | 7 | 8 | 0 | 0 | 0 | 2 | 5

14. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific immunoglobulin M (IgM) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgM responses from circulating lymphocytes. Proportion of children with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom research blood was collected and analyzed. Child Cohort B1 received a single dose of study vaccine and had research blood collected only on Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 0 | 0 | 0 | 0
  LPS | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS: Invaplex
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM (immunoglobulin M) antibody responses to S. sonnei 2a Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine Invaplex-specific IgM responses from circulating lymphocytes. Proportion of children with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 35
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 6 | 11 | 10
Participants | 1 |  | 0 | 1 | 1

16. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS: LPS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM (immunoglobulin M) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- specific IgM responses from circulating lymphocytes. Proportion of children with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 35
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 7 | 11 | 10
Participants | 0 |  | 0 | 1 | 0

17. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS: Invaplex
Description: as for outcome 15
Time Frame: Day 63
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 6 | 10 | 10
Participants | 0 |  | 0 | 0 | 2

18. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS : LPS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM (immunoglobulin M) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS-specific IgM responses from circulating lymphocytes. Proportion of children with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 63
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 6 | 11 | 10
Participants | 0 |  | 0 | 0 | 0

19. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in ALS
Description: The mucosal immune response to WRSS1 was evaluated by assessing specific IgM (immunoglobulin M) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex using the 'antibodies in lymphocyte supernatant' (ALS) assay on culture supernatants of cultured peripheral blood mononuclear cells from different study days before and after vaccination to determine LPS- and Invaplex-specific IgM responses from circulating lymphocytes. Proportion of children with a >= 4-fold increase in antibody titer beyond baseline (mean + 3 standard deviation) was determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: At any time (Day 7 to Day 63)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 2 | 0 | 0 | 1 | 2
  LPS | 0 | 0 | 0 | 1 | 0

20. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgA (immunoglobulin A) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in serum samples at Days -1, 7, 28, 35, 56, 63 and 84. Serotype-speciﬁc LPS from the Walter Reed Army Institute was used to coat the ELISA plates. A ≥4-fold rise in serum antibody titers was considered signiﬁcant. Fold rise is the ratio of follow-up titer/baseline titer. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom research blood was collected and analyzed. Adult Cohort A1 and Child Cohort B1 received a single dose of study vaccine and had research blood collected only on Day 7 and Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 1 | 3 | 2 | 1 | 1 | 0 | 3 | 2
  LPS | 1 | 1 | 3 | 4 | 1 | 0 | 0 | 2 | 3

21. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: Day 28
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  LPS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

22. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: Day 35
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 2 | 0 | 2 |  | 1 | 1 | 3
  LPS | 0 |  | 1 | 0 | 0 |  | 0 | 2 | 5

23. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: Day 56
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 2 | 0 | 1 |  | 0 | 0 | 1
  LPS | 1 |  | 1 | 0 | 0 |  | 0 | 2 | 2

24. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: Day 63
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 7 | 11 | 10
Participants
  Invaplex | 0 |  | 1 | 0 | 1 |  | 0 | 1 | 4
  LPS | 0 |  | 0 | 1 | 2 |  | 2 | 3 | 3

25. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: Day 84
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 3 | 0 | 1 |  | 0 | 1 | 1
  LPS | 0 |  | 0 | 0 | 0 |  | 0 | 0 | 2

26. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Serum
Description: as for outcome 20
Time Frame: At any time (Day 7 to Day 84)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 1 | 7 | 2 | 3 | 1 | 1 | 4 | 6
  LPS | 2 | 1 | 5 | 5 | 3 | 0 | 2 | 5 | 7

27. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgG (immunoglobulin G) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in serum samples at Days -1, 7, 28, 35, 56, 63 and 84. Serotype-speciﬁc LPS from the Walter Reed Army Institute was used to coat the ELISA plates. A ≥4-fold rise in serum antibody titers was considered signiﬁcant. Fold rise is the ratio of follow-up titer/baseline titer. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LPS | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0

28. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: Day 28
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LPS | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2

29. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: Day 35
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 0 | 0 | 0 |  | 0 | 0 | 1
  LPS | 0 |  | 0 | 2 | 0 |  | 0 | 0 | 2

30. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: Day 56
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 1 | 0 | 1 |  | 0 | 0 | 1
  LPS | 0 |  | 0 | 1 | 0 |  | 0 | 0 | 2

31. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: Day 63
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 7 | 11 | 10
Participants
  Invaplex | 0 |  | 1 | 0 | 0 |  | 0 | 0 | 1
  LPS | 0 |  | 0 | 0 | 1 |  | 0 | 0 | 2

32. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: Day 84
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 1 | 0 | 0 |  | 0 | 0 | 0
  LPS | 0 |  | 0 | 0 | 0 |  | 0 | 0 | 2

33. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgG Antibodies in Serum
Description: as for outcome 27
Time Frame: At any time (Day 7 to Day 84)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
  LPS | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 2

34. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in (Immunoglobulin M) IgM Antibodies in Serum
Description: The systemic immune response to WRSS1 was evaluated by assessing the IgM (immunoglobulin M) antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in serum samples at Days -1, 7, 28, 35, 56, 63 and 84. Serotype-speciﬁc LPS from the Walter Reed Army Institute was used to coat the ELISA plates. A ≥4-fold rise in serum antibody titers was considered signiﬁcant. Fold rise is the ratio of follow-up titer/baseline titer. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom research blood was collected and analyzed. Child Cohort B1 received a single dose of study vaccine and had research blood collected only on Day 7 and Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 0 | 0 | 0
  LPS | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: Day 28
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 0 | 0 | 0 | 0 | 0
  LPS | 1 | 0 | 0 | 0 | 1

36. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: Day 35
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 0 | 0 | 0
  LPS | 1 |  | 0 | 0 | 2

37. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: Day 56
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 1 |  | 0 | 0 | 1
  LPS | 0 |  | 0 | 0 | 1

38. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: Day 63
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 7 | 11 | 10
Participants
  Invaplex | 2 |  | 0 | 0 | 0
  LPS | 1 |  | 0 | 0 | 1

39. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: Day 84
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 0 | 0 | 1
  LPS | 2 |  | 0 | 0 | 1

40. Secondary Outcome: Number and Percentage of Child Participants With a 4-fold Rise From Baseline in IgM Antibodies in Serum
Description: as for outcome 34
Time Frame: At any time (Day 7 to Day 84)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 2 | 0 | 0 | 0 | 1
  LPS | 4 | 0 | 0 | 0 | 2

41. Secondary Outcome: Number and Percentage of Adult Participants With a 2-fold Rise From Baseline in IgA and IgG Antibodies in ASC
Description: Antibody Secreting Cell (ASC) by ELISPOT assay responses for IgA (immunoglobulin A) and IgG (immunoglobulin B) ASCs specific for LPS (lipopolysaccharide) and Invaplex were determined at Days -1, 7, 35, and 63. 2-fold increases of LPS and Invaplex specific IgA and IgG in ASC beyond baseline mean + 3 Standard Deviation (SD) were determined. Positive response was ≥8 spots per 1 million peripheral blood mononuclear cells.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom research blood was collected and analyzed. Adult Cohort A1 received a single dose of study vaccine and had research blood collected only on Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3
Number analyzed (Participants) | 9 | 10 | 10 | 8
Participants
  IgA- Invaplex | 2 | 3 | 6 | 3
  IgA- LPS | 4 | 6 | 7 | 6
  IgG- Invaplex | 3 | 4 | 7 | 6
  IgG- LPS | 4 | 2 | 5 | 4

42. Secondary Outcome: Number and Percentage of Adult Participants With a 2-fold Rise From Baseline in IgA and IgG Antibodies in ASC
Description: as for outcome 41
Time Frame: Day 35
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3
Number analyzed (Participants) | 5 | 0 | 10 | 8
Participants
  IgA- Invaplex | 3 |  | 3 | 4
  IgA- LPS | 1 |  | 4 | 3
  IgG- Invaplex | 2 |  | 3 | 5
  IgG- LPS | 2 |  | 1 | 4

43. Secondary Outcome: Number and Percentage of Adult Participants With a 2-fold Rise From Baseline in IgA and IgG Antibodies in ASC
Description: as for outcome 41
Time Frame: Day 63
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3
Number analyzed (Participants) | 6 | 0 | 10 | 8
Participants
  IgA- Invaplex | 2 |  | 3 | 4
  IgA- LPS | 3 |  | 5 | 3
  IgG- Invaplex | 1 |  | 3 | 5
  IgG- LPS | 2 |  | 3 | 4

44. Secondary Outcome: Number and Percentage of Adult Participants With a 2-fold Rise From Baseline in IgA and IgG Antibodies in ASC
Description: as for outcome 41
Time Frame: At any time (Day 7 to Day 63)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3
Number analyzed (Participants) | 9 | 10 | 10 | 8
Participants
  IgA- Invaplex | 5 | 3 | 6 | 6
  IgA- LPS | 5 | 6 | 9 | 6
  IgG- Invaplex | 4 | 4 | 7 | 7
  IgG- LPS | 4 | 2 | 7 | 5

45. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: The mucosal immune response to the WRSS1 was evaluated by assessing Fecal IgA (immunoglobulin A) antibody responses in stool to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in enzyme-linked immunosorbent assay (ELISA) assays, at Days -1, 7, 28, 35, 56, 63, and 84. 4-fold increases of LPS and invaplex-specific IgA in stool beyond baseline mean + 3 SD (standard deviation) were determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer. Pro-inflammatory cytokines (Interleukin 1 beta (IL-1β), Interleukin 8 (IL-8), tumor necrosis factor alpha (TNF-α) and Interferon gamma (IFN-γ)) were measured in stool extracts using commercially available ELISA kits.
Time Frame: Day 7
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom stool was collected and analyzed. Adult Cohort A1 and Child Cohort B1 received a single dose of study vaccine and stool was collected only on Day 7 and Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 3 | 3 | 1 | 2 | 4 | 2 | 4 | 2
  LPS | 1 | 3 | 1 | 2 | 2 | 3 | 2 | 4 | 3

46. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: The mucosal immune response to the WRSS1 was evaluated by assessing Fecal IgA (immunoglobulin A) antibody responses in stool to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in ELISA assays, at Days -1, 7, 28, 35, 56, 63, and 84. 4-fold increases of LPS and invaplex-specific IgA in stool beyond baseline mean + 3 SD (standard deviation) were determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer.Pro-inflammatory cytokines (IL-1β, IL-8, TNF-α and IFN-γ) were measured in stool extracts using commercially available ELISA kits.
Time Frame: Day 28
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 7 | 11 | 10
Participants
  Invaplex | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 3 | 3
  LPS | 2 | 4 | 3 | 2 | 2 | 4 | 2 | 2 | 3

47. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: The mucosal immune response to the WRSS1 was evaluated by assessing Fecal IgA (immunoglobulin A) antibody responses in stool to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in ELISA assays, at Days -1, 7, 28, 35, 56, 63, and 84. 4-fold increases of LPS and invaplex-specific IgA in stool beyond baseline mean + 3 SD (standard deviation) were determined. For those with a zero titer at baseline, fold-rise was defined as the follow-up titer. Pro-inflammatory cytokines (IL-1β, IL-8, TNF-α and IFN-γ) were measured in stool extracts using commercially available ELISA kits.
Time Frame: Day 35
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 2 |  | 1 | 2 | 3 |  | 1 | 2 | 4
  LPS | 2 |  | 1 | 2 | 3 |  | 2 | 3 | 4

48. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: as for outcome 47
Time Frame: Day 56
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 1 |  | 3 | 1 | 1 |  | 0 | 3 | 3
  LPS | 1 |  | 2 | 0 | 2 |  | 1 | 3 | 4

49. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: as for outcome 47
Time Frame: Day 63
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 3 |  | 3 | 2 | 2 |  | 3 | 4 | 3
  LPS | 1 |  | 2 | 0 | 3 |  | 3 | 5 | 3

50. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: as for outcome 47
Time Frame: Day 84
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 2 |  | 1 | 1 | 2 |  | 2 | 4 | 4
  LPS | 1 |  | 2 | 0 | 2 |  | 2 | 5 | 5

51. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in IgA Antibodies in Stool
Description: as for outcome 47
Time Frame: At any time (Day 7 to Day 84)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 5 | 3 | 5 | 5 | 4 | 5 | 5 | 7 | 7
  LPS | 3 | 4 | 5 | 4 | 5 | 4 | 4 | 8 | 7

52. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: Fecal antibody responses were defined as a four-fold rise for specific IgA (immunoglobulin A) or a four-fold rise for the ratio of specific over total IgA at any time point after immunization. Fecal antibody response to the WRSS1 was evaluated by assessing Fecal IgA antibody responses to S. sonnei 2a LPS (lipopolysaccharide) and Invaplex in ELISA assays at Days -1, 7, 28, 35, 56, 63, and 84 . For those participants with a zero titer at baseline fold-rise was defined as the follow-up titer.
Time Frame: Day 7
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 1 | 3 | 0 | 2 | 1 | 2 | 2 | 2 | 3
  LPS | 1 | 4 | 0 | 2 | 1 | 2 | 0 | 3 | 2

53. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: Day 28
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom stool was collected. Participants analyzed (n) were those for whom data was available. Adult Cohort A1 and Child Cohort B1 received a single dose of study vaccine and had stool collected only on Day 7 and Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 7 | 11 | 10
Participants
  Invaplex | 2 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 2
  LPS | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 2

54. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: Day 35
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 0 |  | 0 | 0 | 2 |  | 1 | 2 | 1
  LPS | 0 |  | 0 | 0 | 3 |  | 2 | 2 | 2

55. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: Day 56
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 1 |  | 0 | 0 | 1 |  | 1 | 3 | 0
  LPS | 1 |  | 0 | 0 | 1 |  | 1 | 2 | 0

56. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: Day 63
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 5 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 2 |  | 0 | 0 | 1 |  | 2 | 2 | 1
  LPS | 2 |  | 0 | 0 | 1 |  | 2 | 3 | 1

57. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: Day 84
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 6 | 0 | 10 | 8 | 11 | 0 | 8 | 11 | 10
Participants
  Invaplex | 1 |  | 1 | 0 | 1 |  | 1 | 3 | 2
  LPS | 1 |  | 3 | 0 | 2 |  | 1 | 3 | 4

58. Secondary Outcome: Number and Percentage of Participants With a 4-fold Rise From Baseline in Ratio of Specific IgA to Total IgA Antibodies in Stool
Description: as for outcome 52
Time Frame: At any time (Day 7 to Day 84)
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part B (Children): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 15 | 12 | 8 | 11 | 10
Participants
  Invaplex | 3 | 3 | 1 | 2 | 4 | 2 | 6 | 4 | 4
  LPS | 2 | 4 | 3 | 2 | 4 | 2 | 3 | 5 | 4

59. Secondary Outcome: Number and Percentage of Adult Participants With WRSS1 Shedding at Any Time After Vaccination
Description: Prevalence and distribution of vaccine shedding was determined by quantitative culture and polymerase chain reaction (PCR). The latter measured the mean relative abundance of microbiota by 16S ribosomal ribonucleic acid (rRNA) gene sequence analysis of stool at baseline and post-vaccination days. PCR and stool results were reported as positive if a positive result was reported at any time during the testing period.
Time Frame: At any time (Day 0 to Day 84)
Population: The overall number of participants analyzed (N) were those who received at least one study vaccination and for whom stool was collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Adults): Placebo | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3
Number analyzed (Participants) | 9 | 10 | 10 | 8
Participants | 0 | 1 | 1 | 4

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) and Serious Adverse Event (SAE) data were collected from study Day -1 (inpatient admission day) up to 6 months after any vaccination.
Description: The investigator was responsible for accurate documentation of all AEs and SAEs. The Principal Investigator monitored all AEs until Day 168 (for cohort A1 and B1) and Day 224 (for cohort A2, A3, B2 B3 and B4). All SAEs were followed up until the event resolved or stabilized or the participant was lost to follow-up. Continued follow-up was at the discretion of the PI based on good clinical management or until the participant was referred to another institution for continued care.
Arm/Group | Part A (Adults): Cohort A1 | Part A (Adults): Cohort A2 | Part A (Adults): Cohort A3 | Part A (Adults): Placebo | Part B (Children): Cohort B1 | Part B (Children): Cohort B2 | Part B (Children): Cohort B3 | Part B (Children): Cohort B4 | Part B (Children): Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9 | 0/12 | 0/12 | 0/12 | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10 | 0/9 | 1/12 | 0/12 | 0/12 | 1/12 | 1/16
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 8/10 | 6/9 | 10/12 | 9/12 | 9/12 | 12/12 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Adults): Cohort A1 (N=10) | Part A (Adults): Cohort A2 (N=10) | Part A (Adults): Cohort A3 (N=10) | Part A (Adults): Placebo (N=9) | Part B (Children): Cohort B1 (N=12) | Part B (Children): Cohort B2 (N=12) | Part B (Children): Cohort B3 (N=12) | Part B (Children): Cohort B4 (N=12) | Part B (Children): Placebo (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Voluntary abortion
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Adults): Cohort A1 (N=10) | Part A (Adults): Cohort A2 (N=10) | Part A (Adults): Cohort A3 (N=10) | Part A (Adults): Placebo (N=9) | Part B (Children): Cohort B1 (N=12) | Part B (Children): Cohort B2 (N=12) | Part B (Children): Cohort B3 (N=12) | Part B (Children): Cohort B4 (N=12) | Part B (Children): Placebo (N=16)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 5 (7) | 2 (2)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (9) | 3 (3) | 3 (3) | 2 (2)
Conjunctivitis allergic (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection parasitic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 7 (8) | 4 (4) | 6 (7) | 2 (2) | 6 (7)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abrasion injury
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 5 (6) | 2 (3)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Abrasion
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No